CLINICAL TRIAL: NCT06919666
Title: Phase Ib/II Study of NT219 in Combination With Pembrolizumab or Cetuximab in Patients With Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma (HNSCC)
Brief Title: NT219 Combined With Standard of Care Biologic Therapy in Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Purple Biotech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 24-0689.cc
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Head and Neck Cancer; Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 NT219 plus pembrolizumab (Experimental): Cohort 1 will enroll patients who have not received PD-1 inhibition in the relapsed/metastatic setting or have received and derived significant clinical benefit from PD-1 inhibition as their first line of therapy. Patients will be treated with NT219 75 mg/kg IV once weekly plus pembrolizumab 200 mg once every three weeks. The first 6 patients will be required to clear a DLT window of 21 days as an abbreviated safety lead-in.
  Interventions: Drug: NT219
- Cohort 2 NT219 plus cetuximab (Experimental): Cohort 2 will enroll patients who had progression of disease without clinical benefit from PD-1 inhibition or have received ≥2 prior lines of therapy and are good candidates for cetuximab. Patients will be treated with NT219 75mg/kg IV once weekly plus cetuximab given as an initial loading dose of 400 mg/m2 followed by maintenance dosing of 250 mg/m2 once weekly.
  Interventions: Drug: NT219

INTERVENTIONS:
Drug: NT219 — NT219 is a first-in-class small molecule targeting IRS 1/2 and STAT3. Preclinical studies in melanoma have shown NT219 induces PD-L1 expression in vitro and in vivo, resulting in increased efficacy of PD-1 inhibition via synergistic antitumor effect in PD-1 sensitive models and restoration of sensitivity in resistant models. NT219 also synergized with cetuximab in vitro and reversed cetuximab resistance in a head and neck cancer xenograft platform.

SUMMARY:
Fixed dose NT219 weekly plus pembrolizumab every 3 weeks or cetuximab weekly to be continued until progression, unacceptable toxicity, or investigator or participant decision.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and over.
* ECOG PS 0-2.
* Incurable head and neck squamous cell carcinoma of mucosal origin (oral cavity, tongue, oropharynx, pharynx, larynx, sinonasal and non-EBV-driven NPC).
* Adequate organ and marrow function as defined by routine lab testing including calculated creatinine clearance >60 mL/min, total bilirubin < 1.5x the ULN, ALT and AST <5x the ULN, ANC >1500, and platelets >100,000.
* Measurable disease by RECIST on CT (including a diagnostic CT performed as part of a PET-CT) or MRI available for review.
* Recovered from clinically significant adverse events of most recent anti-cancer therapy prior to enrollment.
* Cohort 1: In addition to the general inclusion criterion, patients with tumor tissue CPS >1 for whom single agent pembrolizumab is appropriate OR who derived significant clinical benefit from anti-PD-1 therapy (as single agent or combination) in the first line setting. No more than 7 patients with each profile (PD-1 inhibitor naïve vs PD-1 inhibitor experienced with benefit) can be enrolled in the first stage of Cohort 1.

  o Significant clinical benefit is defined as treatment duration >=6 months and/or PR/CR as best objective response prior to disease progression.
* Cohort 1: In addition to the above inclusion criterion, patients must have accessible sites of disease not involving target lesions that are amenable to sequential biopsies, and participants willing to undergo sequential tumor biopsies as long as the treating investigator considers to be clinically safe.
* Cohort 2: In addition to the general inclusion criteria, patients have had progression or recurrence in the relapsed/metastatic setting to PD-1 inhibitors given with or without cytotoxic chemotherapy without significant clinical benefit OR who are candidates for cetuximab monotherapy.

  * Significant clinical benefit is defined as treatment duration >=6 months and/or PR/CR as best objective response prior to disease progression.

Exclusion Criteria:

* Unknown origin squamous cancer.
* EBV-driven NPC.
* 4 lines or more in the relapsed/metastatic setting.
* Pregnant or lactating, as the effects of NT219 on a fetus or child are unknown. Patients who are capable of childbearing or have partners capable of childbearing must use two forms of birth control including a barrier method to avoid pregnancy.
* Known central nervous system metastases unless previously treated and clinically stable for at least one month.
* Major surgery within 4 weeks or minor surgery within 1 week of starting therapy.
* Known active HIV infection, unless treated with no detectable virus, or active HIV infection based on screening testing.
* Participants with chronic hepatitis B virus (HBV) infection with active disease that meets the criteria for anti-HBV therapy and are not on suppressive antiviral therapy for at least 4 weeks prior to the first dose of study treatment.
* Patients with known hepatitis C virus (HCV) who have not completed curative antiviral treatment at least 4 weeks prior to first dose of study treatment or have an HCV viral load above the limit of quantification at screening.
* Prior anti-cancer biologic agent within 4 weeks prior to Study Day 1, or prior chemotherapy, targeted small molecular therapy, or radiation therapy within 2 weeks prior to Study Day 1, as wash-out considerations.
* Vaccine administration within 4 weeks before the first dose of NT219
* Serious systemic infection within 4 weeks of the first dose of the study treatment, or clinically significant infection requiring hospitalization and/or IV anti-infective therapy within 2 weeks of the first dose of the study treatment.
* Receipt of any organ transplantation including autologous and allogeneic stem cell transplantation, with the exception of transplants that do not require immunosuppression.
* Diagnosed and/or treated for any other additional malignancy within 2 years of the first dose of study treatment with the exception of curatively treated basal cell or squamous cell carcinoma of the skin and curatively resected in situ cancers. Other exceptions may be considered with the PI's consultation.
* Cohort 1: In addition to the general exclusion criteria, patients with active autoimmune disease requiring systemic treatment in the past two years with use of disease modifying agents, corticosteroids, or immunosuppressive drugs. Replacement therapy such as thyroxine, insulin, or physiologic corticosteroids is allowed. Well-managed or inactive autoimmune disorders, such as Hashimoto's thyroiditis, are allowed at the discretion of the PI.
* Cohort 1: Any condition requiring systemic treatment with >10mg prednisone or equivalent corticosteroid daily or other systemic immunosuppressive medication within 2 weeks of the first dose of study treatment. Topical, intranasal, intrabronchial, and ocular steroids are allowed. Steroids used as premedication for allergic reactions or as prophylactic management of AEs related to the study drugs specific in this protocol are allowed.
* Cohort 2: Any of the following within 6 months of starting study treatment: ST elevation myocardial infarction, severe or unstable angina, uncontrolled cardiac ventricular arrhythmia, coronary or peripheral artery bypass graph or stent, cerebrovascular accident or stroke, or severe/uncontrolled congestive heart failure. Deep vein thrombosis that are hemodynamically stable do not exclude enrollment if the patient has been on a stable dose of anticoagulant for at least three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2030-02 (Estimated); Study Completion 2031-02 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate following treatment with NT219 plus pembrolizumab (cohort 1) or cetuximab (cohort 2). | Tumor assessments will be completed every 9 weeks from enrollment/baseline until the final study visit. Additional imaging can occur at 60 days post-treatment +/- 7 days at the discretion of the investigator.
  Objective response rate is defined as the percentage of participants who have confirmed best response of complete response or partial response as determined by the investigator. Response will be assessed by RECIST 1.1 or iRECIST (when applicable, cohort 1 only) at baseline (within 28 days of C1D1) and every 9 weeks +/- 10 days while on treatment. All scans during study intervention will be repeated using the same method (CT, PET-CT, or MRI).

SECONDARY OUTCOMES:
Rate of occurence of dose-limiting toxicity (DLT) within the first 21-day cycle of NT219 plus pembrolizumab (Cohort 1 only) | DLTs will be collected from C1D1 to C1D21 of NT219 plus pembrolizumab
  DLT is defined as any of the following occuring during Cycle 1 of NT219 administered in combination with pembrolizumab: Grade >=3 non-hematologic toxicity, Grade >=4 neutropenia >7 days, Grade >=3 thrombocytopenia with clinically significant bleeding, neutropenic fever, any Hy's law case (AST or ALT >3 x ULN AND total bilirubin >2x ULN AND alk phos <2x ULN AND no other reason for liver injury), and any death not clearly due to underlying disease or extraneous causes. The following Grade >=3 non-hematologic toxicities are NOT considered DLTs: Grade 3 nausea, vomiting, or diarrhea <72 hours with adequate antiemetic and other supportive care; Grade 3 fatigue lasting <7 days; Grade >=3 or higher electrolyte abnormalities lasting up to 72 hours which are not clinically complicated and resolve spontaneously or respond to conventional medical interventions; Grade 3 amylase or lipase elevation not associated with symptoms or clinical manifestations of pancreatitis.
Occurence of treatment-emergent and treatment-related adverse events (AEs) in patients treated with NT219 plus pembrolizumab (cohort 1) or cetuximab (cohort 2). | AEs will be collected from C1D1 until the final study visit
  AEs will be graded according to NCI CTCAE v5.0.
Progression-free survival (PFS) in patients treated with NT219 plus pembrolizumab (Cohort 1) or cetuximab (Cohort 2) | First dose of NT219 plus pembrolizumab (Cohort 1) or cetuximab (Cohort 2) until progressive disease, death, or loss of follow-up.
  PFS is defined as the time from first dose of NT219 plus pembrolizumab (Cohort 1) or cetuximab (Cohort 2) until investigator-assessed radiographic progressive disease, death, or loss of follow-up, whichever occurs first.
Overall survival in patients treated with NT219 plus pembrolizumab (Cohort 1) or cetuximab (Cohort 2) | First dose of NT219 plus pembrolizumab (Cohort 1) or cetuximab (Cohort 2) until death or loss of follow-up.
  Overall survival is defined as the time from first dose of NT219 plus pembrolizumab (Cohort 1) or cetuximab (Cohort 2) until death or loss of follow-up, whichever occurs first.
Duration of response in patients treated with NT219 plus pembrolizumab (Cohort 1) or cetuximab (Cohort 2) | Time from response to NT219 plus pembrolizumab (Cohort 1) or cetuximab (Cohort 2) to progression, death, or loss of clinical follow-up.
  Duration of response is defined as the time from response to NT219 plus pembrolizumab (Cohort 1) or cetuximab (Cohort 2) to progression, death, or loss of clinical follow-up, whichever occurs first.
Clinical benefit rate for patients treated with NT219 plus pembrolizumab (Cohort 1) or cetuximab (Cohort 2) | Tumor assessments will be completed every 9 weeks from enrollment/baseline until the final study visit. Additional imaging can occur at 60 days post-treatment +/- 7 days at the discretion of the investigator.
  Clinical benefit rate is defined as the percentage of participants who have confirmed best response of complete response, partial response, or stable disease as determined by the investigator according to RECIST or iRECIST (when applicable, Cohort 1 only).

OTHER OUTCOMES:
Change from Baseline in Tumor Expression of Immune Biomarkers in patients treated with NT219 plus pembrolizumab (Cohort 1 only) | Baseline tumor tissue collection will occur during the screening window, post-treatment tumor tissue will be collected at C2D8 +/- 2 days
  Baseline and post-treatment tumor tissue will be collected and analyzed for expression of immune biomarkers using immunohistochemistry
Change from Baseline in Immune Cell Profiles in tumor tissue from patients treated with NT219 plus pembrolizumab (Cohort 1 only) | Baseline tumor tissue collection will occur during the screening window, post-treatment tumor tissue will be collected at C2D8 +/- 2 days
  Baseline and post-treatment tumor tissue will be collected and analyzed for immune cell profiles in tumor and surrounding tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Alice Weaver, MD, PhD, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - Universtiy of Colorado Hospital, Aurora, Colorado
  - UCHealth Highlands Ranch Hospital, Highlands Ranch, Colorado